CLINICAL TRIAL: NCT06896604
Title: Comparison of the Effects of Low-Flow and High-Flow Desflurane Anesthesia on Optic Nerve Sheath Diameter in Laparoscopic Cholecystectomy Surgeries
Brief Title: Changes in Optic Nerve Sheath Diameter in Desflurane Based General Anesthesia During Laparoscopic Cholecystectomies
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mervenur Gizem Öztürk, resident doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMTRH-AR-MGO-01
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: Low Fresh Gas Flow, Desflurane; Desflurane; Cholecystectomy, Laparoscopic; Spectroscopy, Near-Infrared; Optic Nerve Sheath Diameter Sonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low flow anesthesia with desflurane: After standard induction procedures, the fresh gas flow was reduced to 1 L/min during the maintenance phase of inhalation anesthesia with desflurane.
  Interventions: Device: Ocular Ultrasonography for measuring Optic Nerve Sheath Diameter
- high flow anesthesia with desflurane: After standard induction procedures, the fresh gas flow was set to 3 L/min during the maintenance phase of inhalation anesthesia with desflurane.
  Interventions: Device: Ocular Ultrasonography for measuring Optic Nerve Sheath Diameter

INTERVENTIONS:
Device: Ocular Ultrasonography for measuring Optic Nerve Sheath Diameter — In the study, the investigators measured the optic nerve sheath diameter to observe its effects on intracranial pressure and used ocular ultrasonography for this measurement.

SUMMARY:
In this study, the investigators to observe the effects of different fresh gas flow rates, which are frequently used in general anesthesia practice, on optic nerve sheath diameter during laparoscopic cholecystectomy surgeries under general anesthesia with desflurane.

DETAILED DESCRIPTION:
All inhalational anesthetic agents, particularly desflurane, have direct vasodilatory effects on cerebral vessels under normocapnic and normotensive conditions. In a dose-dependent manner, they lead to a moderate increase in cerebral blood flow (CBF) and intracranial pressure (ICP). Except for patients with high ICP due to mass lesions or head trauma, these changes in CBF are generally well tolerated in most patients undergoing general anesthesia. To prevent complications such as hypoxia, hypercapnia, and hemodynamic changes that may arise due to the anesthetic agent's dosage, strict intraoperative monitoring and follow-up are required. Advances in monitoring and anesthesia devices allow for the measurement of respiratory and hemodynamic parameters, as well as inhaled and exhaled gas concentrations, facilitating the assessment of cerebral perfusion and ICP using ultrasonography.

Intracranial pressure may increase independently of anesthetic agents and techniques due to patient positioning during surgery or pneumoperitoneum in laparoscopic procedures. Near-infrared spectroscopy (NIRS) measures regional cerebral oxygen saturation, enabling early detection of potential changes in cerebral perfusion and oxygenation during surgical procedures under anesthesia. Additionally, ultrasound-guided optic nerve sheath diameter (ONSD) measurement is a non-invasive, easily applicable, cost-effective, and reproducible technique for evaluating ICP changes.

In this study, the investigators to investigate the effects of different fresh gas flow rates, which are frequently used in general anesthesia practice, on ONSD during laparoscopic cholecystectomy procedures under general anesthesia with desflurane.

After obtaining approval from the ethics committee, patients aged 18-65 years, classified as American Society of Anesthesiologists (ASA) physical risk score I-III, who are scheduled for elective laparoscopic cholecystectomy under general anesthesia at Fatih Sultan Mehmet Training and Research Hospital, will be included in the study. Based on a power analysis conducted using the G*Power program, it was determined that a minimum of 44 patients would be required for 90% power, and the study plans to include 60 patients. Prior to the surgery, patients will be informed about the study, and their consent will be obtained. Measurements of optic nerve sheath diameter (ONSD) using ultrasonography (USG) will be performed on patients before the surgery, during the surgery, and after the surgery. The measurements will be conducted by the anesthesia team, will not be reflected as a service in the patient's medical file, and no fees will be charged to the patient or the institution. Independently from the study team, the anesthesiologist will classify patients into two observational subgroups based on their choice of fresh gas flow rates during desflurane anesthesia: Group I will consist of patients with a fresh gas flow rate of 1 L/min, and Group II will consist of patients with a fresh gas flow rate of 3 L/min.

Patients admitted to the operating room will undergo standard monitoring, including electrocardiogram (ECG), non-invasive blood pressure monitoring, peripheral oxygen saturation (SpO2) monitoring, body temperature measurement (via temporal artery surface temperature measurement using the 3M Spot ON method), bispectral index (BIS) monitoring for anesthesia depth, and near-infrared spectroscopy (NIRS) monitoring for cerebral perfusion. Following this, ONSD measurements will be made on both the right and left eyelids using USG in patients without premedication. The average of two measurements taken from each eye will be recorded. After completion of measurements, standard preoxygenation (3 minutes with a 100% oxygen mask) will be followed by intravenous (IV) induction with 2-2.5 mg/kg propofol, 2 mcg/kg fentanyl, and 0.6 mg/kg rocuronium. After sufficient muscle relaxation, patients will be orotracheally intubated, and mechanical ventilation will be provided with end-tidal CO2 (EtCO2) maintained within normal limits (35-40 mmHg). Anesthesia maintenance will be provided using a 50% O2-Air mixture with 4-6% desflurane at the fresh gas flow rates preferred by the anesthesiologists, either 1 L/min or 3 L/min. Intraoperative analgesia will be maintained with an IV remifentanil infusion of 0.05-0.2 mcg/kg/min. Anesthetic drugs will be titrated to maintain BIS values between 40-60, and NIRS measurements will ensure that the cerebral oxygenation does not decrease by more than 20% from the baseline. Heart rate (HR) and/or mean arterial pressure (MAP) will also be adjusted to remain within 20% of the baseline. Pneumoperitoneum pressure will be maintained at a standard value of 14 mmHg during surgery. After cholecystectomy, postoperative analgesia will be provided with 1g of paracetamol and 1 mg/kg tramadol, and postoperative nausea prophylaxis will be achieved with 4 mg of ondansetron IV. At the end of the surgery, in patients with spontaneous respiratory effort, neuromuscular blockade will be reversed with 2 mg/kg sugammadex IV. Once sufficient respiratory effort and BIS ≥85 are observed, patients will be extubated and transferred to the recovery unit once they are conscious, with restored muscle strength and hemodynamically stable. During the operation, routine hemodynamic parameters, including SpO2, non-invasive arterial pressure, heart rate, respiratory rate, body temperature, EtCO2, inspiratory-expiratory oxygen and anesthetic gas concentrations, airway pressures (Ppeak, Pplateau), NIRS, and BIS values will be monitored and recorded simultaneously. ONSD measurements will be performed pre-anesthesia (T0), post-intubation (T1), at the 5th minute following pneumoperitoneum (T2), at the 20th minute after pneumoperitoneum (T3), after desufflation (T4), and at 15 minutes postoperatively in the recovery unit (T5), and will be recorded. Additionally, nausea, vomiting, and shivering occurrences will be noted in the recovery phase. Patients with an Aldrete score of ≥8 will be transferred to the ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients Undergoing Elective Laparoscopic Cholecystectomy Under General Anesthesia
* Patients aged 18-65 years with an American Society of Anesthesiologists (ASA) physical status classification of I-III and a body mass index (BMI) < 35 kg/m²
* Patients who have provided informed consent

Exclusion Criteria:

* Patients under 18 or over 65 years old, those classified as ASA IV-V, or with a BMI ≥ 35 kg/m²
* Patients with conditions that may lead to increased intracranial pressure (e.g., intracranial mass, aneurysm, head trauma), a history of intracranial surgery, previous ischemic or hemorrhagic stroke, or neurological diseases
* Patients with a history of glaucoma or cataract surgery
* Patients undergoing emergency surgical procedures
* Patients with severe cardiac, renal, pulmonary, or hepatic failure
* Patients who do not provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years with an American Society of Anesthesiologists (ASA) physical status classification of I-III and a body mass index (BMI) < 35 kg/m², undergoing elective laparoscopic cholecystectomy under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Measurement of Optic Nerve Sheath Diameter for Observing Intracranial Pressure Increase | through study completion, an average of 2 months
  Investigation of the Effects of Desflurane Administration with Different Fresh Gas Flow Rates on Optic Nerve Sheath Diameter

SECONDARY OUTCOMES:
Monitoring Cerebral Perfusion Using Near-Infrared Spectroscopy | through study completion, an average of 2 months
  Comparison of the Effects of Different Fresh Gas Flow Rates on Cerebral Perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Oznur Demiroluk, As Prof, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Geeraerts T, Merceron S, Benhamou D, Vigue B, Duranteau J. Non-invasive assessment of intracranial pressure using ocular sonography in neurocritical care patients. Intensive Care Med. 2008 Nov;34(11):2062-7. doi: 10.1007/s00134-008-1149-x. Epub 2008 May 29. PMID 18509619
- [Result] Akbas S, Ozkan AS. Comparison of effects of low-flow and normal-flow anesthesia on cerebral oxygenation and bispectral index in morbidly obese patients undergoing laparoscopic sleeve gastrectomy: a prospective, randomized clinical trial. Wideochir Inne Tech Maloinwazyjne. 2019 Jan;14(1):19-26. doi: 10.5114/wiitm.2018.77265. Epub 2018 Jul 24. PMID 30766625
- [Result] Choi ES, Jeon YT, Sohn HM, Kim DW, Choi SJ, In CB. Comparison of the effects of desflurane and total intravenous anesthesia on the optic nerve sheath diameter in robot assisted laparoscopic radical prostatectomy: A randomized controlled trial. Medicine (Baltimore). 2018 Oct;97(41):e12772. doi: 10.1097/MD.0000000000012772. PMID 30313092
- [Result] Oterkus M, Donmez I, Nadir AH, Rencuzogullari I, Karabag Y, Binnetoglu K. The effect of low flow anesthesia on hemodynamic and peripheral oxygenation parameters in obesity surgery. Saudi Med J. 2021 Mar;42(3):264-269. doi: 10.15537/smj.2021.42.3.20200575. PMID 33632904
- [Result] Tekin EA, Gultop F, Baskurt NA. Minimal and normal-flow general anesthesia in patients undergoing surgery in prone position: impact on hemodynamics and regional cerebral oxygenation. Acta Cir Bras. 2023 Mar 24;38:e380523. doi: 10.1590/acb380523. eCollection 2023. PMID 36995818
- [Result] Bingol Tanriverdi T, Tercan M, Gusun Halitoglu A, Kaya A, Patmano G. Comparison of the Effects of Low-flow and Normal-flow Desflurane Anaesthesia on Inflammatory Parameters in Patients Undergoing Laparoscopic Cholecystectomy. Turk J Anaesthesiol Reanim. 2021 Feb;49(1):18-24. doi: 10.5152/TJAR.2020.30. Epub 2020 Nov 30. PMID 33718901
- [Result] Bedforth NM, Hardman JG, Nathanson MH. Cerebral hemodynamic response to the introduction of desflurane: A comparison with sevoflurane. Anesth Analg. 2000 Jul;91(1):152-5. doi: 10.1097/00000539-200007000-00028. PMID 10866903
- [Result] Jiang Z, Wu Y, Liang F, Jian M, Liu H, Mei H, Han R. Brain relaxation using desflurane anesthesia and total intravenous anesthesia in patients undergoing craniotomy for supratentorial tumors: a randomized controlled study. BMC Anesthesiol. 2023 Jan 10;23(1):15. doi: 10.1186/s12871-023-01970-z. PMID 36624384